CLINICAL TRIAL: NCT06108349
Title: A Randomized Controlled Trial of Topical Cannabidiol for the Treatment of Carpal Tunnel Syndrome
Brief Title: Topical Cannabidiol for Treating Carpal Tunnel Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Brent DeGeorge, Plastic Surgeon and Assistant Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HSR230375
Record Dates: First submitted 2023-10-04; First posted 2023-10-31 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Distal median nerve compression; Entrapment neuropathy
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy; Charcot-Marie-Tooth Disease | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Experimental): Participants will receive 5mL syringe with Cannabidiol (Investigational drug) in it.
  Interventions: Drug: Cannabidiol
- Placebo (No Intervention): Participants will receive 5mL syringe with Shea Butter cream (Placebo) in it.

INTERVENTIONS:
Drug: Cannabidiol — Cannabidiol (CBD) is a non-psychoactive minor cannabinoid component of Cannabis sativa that is emerging as a treatment to mitigate pain, numbness, and tingling associated with peripheral neuropathy. CBD acts through multiple receptors to modulate central and peripheral neuropathic signaling pathways to alleviate pain.
  Arms: Cannabidiol

SUMMARY:
The Purpose of this study is to assess the safety and efficacy of Cannabidiol on treatment of Carpal Tunnel Syndrome.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS), or compression neuropathy of the median nerve at the wrist, is the most common entrapment neuropathy affecting up to 15% of the general population Non-operative interventions for CTS include night-time splinting, physical therapy, and corticosteroid administration, however only surgery is considered a definitive treatment for CTS. There is an unmet need for novel, effective non-operative options for the treatment of CTS to provide care for patients who cannot undergo surgery for medical reasons or do not feel comfortable proceeding with a surgical option.

Cannabidiol (CBD) is a non-psychoactive minor cannabinoid component of Cannabis sativa that is emerging as a treatment to mitigate pain, numbness, and tingling associated with peripheral neuropathy. Pre-clinical data indicates that CBD acts through multiple receptors to modulate central and peripheral neuropathic signaling pathways to alleviate pain - specifically in pre-clinical models of compression neuropathy as in CTS. This pilot trial seeks to investigate whether CBD is a safe, feasible, and effective treatment for CTS in patients with confirmed mild to moderate CTS receiving standardized physiotherapy with primary endpoints assessing feasibility, symptom severity, and/or disability and also highlights the gap in knowledge regarding the clinical utility of cannabinoids

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18 years or older.
4. Females of childbearing potential must have a negative urine and blood pregnancy test at Screening and a negative urine pregnancy test before study drug is administered. Females must abstain from sex or use a highly effective method of contraception during the period from Screening to administration of study drug and for 30 days after the last dose of study medication. Standard acceptable methods include abstinence or the use of a highly effective method of contraception, including; hormonal contraception, diaphragm, cervical cap, vaginal sponge, condom with spermicide, vasectomy, intrauterine device. If females are of non-child bearing potential, they must be post-menopausal defined as: age > 55 with no menses within the past 12 months, or history of hysterectomy, or history of bilateral oophorectomy, or bilateral tubal ligation.
5. Males must consent to use a medically acceptable method of contraception throughout the entire study period and for 90 days after their last study drug application. They must agree to not donate sperm for 90 days after their last study drug application.
6. Presence of clinical diagnosis of carpal tunnel syndrome with a CTS-6 score greater than 12 who have undergone electrodiagnostic testing with mild to moderate carpal tunnel syndrome

Exclusion Criteria:

1. Subject does not speak English.
2. Subject is blind.
3. Severe cardiac, pulmonary, liver and /or renal disease.
4. Coumadin use at time of screening.
5. History of mental illness.
6. Subjects who are incarcerated.
7. History of drug or substance abuse.
8. Pre-existing CBD or hemp based product usage.
9. Prior carpal tunnel release surgery or carpal tunnel corticosteroid injection ≤ 6 months prior.
10. History of constant, unremitting numbness or tingling.
11. History of thenar atrophy.
12. Patients with severe changes on electrodiagnostic testing.
13. Patients with a concomitant diagnosis of cervical radiculopathy, peripheral neuropathy, cubital tunnel syndrome, fibromyalgia, chronic regional pain syndrome, or other upper extremity neuropathy
14. Females who are pregnant, nursing or planning a pregnancy; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception as outlined in this protocol from Screening to the first dose of study medication and for 30 days after the last dose of study medication. Standard acceptable methods include abstinence or the use of a highly effective method of contraception, including; hormonal contraception, diaphragm, cervical cap, vaginal sponge, condom with spermicide, vasectomy, intrauterine device.
15. Any skin disease or condition, including eczema, psoriasis, melanoma, acne or contact dermatitis, scarring, imperfections, lesions, tattoos or discoloration that may affect treatment application, application site assessments, or affect absorption of the study drug.
16. Subjects taking prescription or non-prescription medication which are substrates of CYP3A4 (Itraconazole, Ketoconazole, Azamulin, Troleandomycin, Verapamil, John's wart, Phenobarbital), CYP2C19 (Nootkatone, Ticlopidine, Rifampin, Omeprazole), CYP2C8 (Montelukast, Quercetin, Phenelzine, Rifampin, Clopidogrel) , CYP2C9 (Sulfaphenazole, Tienilic acid, Carbamazepine, Apalutamide, Fluconazole, Celecoxib), CYP1A2 (alpha-Naphthoflavone, Furafylline, Phenytoin, Rifampin, Ritonavir, smoking, Teriflunomide, Ciproflaoxacin, oral contraceptives, Alloprinol) and CYP2B6 (Sertraline, Phencyclidine, Thiotepa, Ticlopidine, Carbamazepine, Efavirenez, Rifampin, Bupropion) within 14 days of the study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of CBD as a topical treatment for CTS is determined by the investigator by evaluating the Recruitment Rate, medication compliance rate and retention rate. | 2 weeks and then crossover to other cream for 2 more weeks after a 1 week washout period.
  1. The Study PI uses recruitment materials and participant materials for enrolling the subjects.
     study participants will be randomized to either the treatment group or placebo group (1:1 ratio) once consent is signed and inclusion/exclusion criteria are satisfied. Recruitment rate is calculated by comparing number of patients with CTS willing to undergo randomization compared to patients offered enrollment in the trial.
  2. Study medication will be dispensed to the subjects by the study team and are returned to the study team at the next visit. study drug accountability will be maintained by the research team.
  3. Retention Rate will be calculated by number of patients completing the follow up visit. The investigator or designee will make every effort to regain contact with the participant.

SECONDARY OUTCOMES:
The efficacy of CBD as a topical treatment for carpal tunnel syndrome is measured by a. Change in symptom severity as reported with the Boston Carpal Tunnel Symptom Severity Scale from baseline and study Days 14, 21 and 28. | 2 weeks
  The Boston Carpal Tunnel Score is a patient-reported questionnaire that examines symptom severity and overall functional status of patients with carpal tunnel syndrome. The Symptom Severity Scale (SSS) with 11 questions is scored on a Likert scale of 1-5 and the Functional Status Scale (FSS) with 8 questions is scored from 1-5 with 1 as no difficulty and 5 as difficult from Baseline and Study Days 14, 21 and 28.
The efficacy of CBD as a topical treatment for carpal tunnel syndrome is measured by change in patient reported outcomes measured by SANE scores from baseline and study Days 14, 21 and 28. | 2 weeks
  SANE Score: Single Assessment Numerical Evaluation (SANE) is a validated metric for musculoskeletal pain which can be applied to any joint or region of interest. This assessment will be performed at Baseline and Study Days 14, 21 and 28. The physician will ask the subject each question and record the response on the source document.
The efficacy of CBD as a topical treatment for carpal tunnel syndrome is measured by change in Patient reported outcomes measurement information system from baseline and study Days 14, 21 and 28. | 2 weeks
  The PROMIS 10 consists of ten (10) items that measure physical health, physical functioning, general mental health, emotional distress, satisfaction with social activities and relationships, ability to carry out usual social activities and roles, pain, fatigue and overall quality of life.
The efficacy of CBD as a topical treatment for carpal tunnel syndrome is measured by change in VAS scores from baseline and study Days 14, 21 and 28. | 2 weeks
  VAS Scores: The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
  It is assessed from baseline and study Days 14, 21 and 28.
Along with efficacy, safety of CBD is measured by performing set of Laboratory tests | 2 weeks
  Laboratory Testing: At Screening a blood draw will be performed on all female subjects of childbearing age. The following tests will be ordered:
  * Pregnancy Testing (if applicable) (Screening only)
  * Urine Pregnancy Test (if applicable) (Screening and Day 0 before dosing only)
Safety of CBD is measured by collecting relevant Medical History as a part of safety assessment. | 2 weeks
  Medical History: Relevant medical history, including history of mental illness, drug or substance abuse, history of hemp-based product usage and other pertinent history will be recorded in the case report form.
Safety of CBD is measured by performing skin monitoring tests and physical examination. | 2 weeks
  Investigator will assess the CBD cream site for adverse events at baseline and at every subsequent visit.
  A score will be given corresponding to the assessment tool.
  If the score is "0"- No erythema If the score is "1"- Minimal erythema If the score is "2"- Moderate erythema with sharply defined borders If the score is "3"- Intense erythema with or without edema If the score is "4"- Intense erythema with edema and blistering/erosion